CLINICAL TRIAL: NCT05302804
Title: The Influence of Topical Menthol Gel on Thermoregulatory and Perceptual Outcomes During Exercise Within the Heat
Brief Title: The Influence of Menthol Gel During Exercise With Heat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0111-22-FB
Record Dates: First submitted 2022-03-17; First posted 2022-03-31 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Acute Exercise; Heat Exposure
Keywords: heat exposure; menthol; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Each Subject acts as their own control in a repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Menthol Gel first, then hypoallergenic gel (Experimental): Participants randomized to receive menthol gel first then hypoallergenic gel after 7 day washout.
  Gel is applied to the skin (arm and thigh). Participants walk on a treadmill for 30 minutes (3.5 mph at 5% grade) in 38°C and 60% relative humidity.
  Interventions: Drug: Menthol Gel; Drug: Control Gel
- Hypoallergenic Gel first, then menthol (Experimental): Participants randomized to receive hypoallergenic gel first then menthol gel after 7 day washout.
  Gel is applied to the skin (arm and thigh). Participants walk on a treadmill for 30 minutes (3.5 mph at 5% grade) in 38°C and 60% relative humidity.
  Interventions: Drug: Menthol Gel; Drug: Control Gel

INTERVENTIONS:
Drug: Menthol Gel — 5% menthol gel applied from shoulder to wrist and mid thigh to ankle, 30 minute treadmill walk (3.5 mph at 5% grade at 38°C, 60% relative humidity)
  Other Names: BioFreeze
Drug: Control Gel — Hypoallergenic gel applied from shoulder to wrist and mid thigh to ankle, 30 minute treadmill walk (3.5 mph at 5% grade at 38°C, 60% relative humidity)
  Other Names: placebo

SUMMARY:
The purpose of this study is to examine the human thermoregulatory impact of applying a commercially available menthol gel (BioFreeze) to the skin prior to moderate intensity walking under heated conditions. Experimental Visits will consist of 30 min of treadmill walking at a moderate pace (3.5 mph, 5% grade) under hot conditions (38°C, 60%RH) and will be randomized and counterbalanced for BioFreeze or a hypoallergenic gel (control) application. Gels will be applied to areas commonly exposed during outdoor activity in warm conditions (shoulder to wrist, mid thigh to ankle). Accordingly, participants will wear shorts and a tank top shirt during exercise. Core temperature, skin temperature, galvanic skin response, laser doppler blood flow, and heart rate will be continuously recorded throughout the exercise bout via an integrated analog to digital converter. Sweat will be collected during exercise using commercially available absorbent patches. Thermal sensation will be assessed throughout exercise via the American Society of Heating, Refrigerating and Air-Conditioning Engineers (ASHRAE) thermal sensation likert scale (cold to hot). Lastly, nude body weight will be recorded pre and post exercise for sweat rate determination. The BioFreeze and control trials will be separated by a 7-14 day washout period.

DETAILED DESCRIPTION:
3 experimental visits to the laboratory will be conducted. All visits will take place at the University of Nebraska at Omaha, Exercise Physiology Laboratory. Visit 1 will consist of the physical activity readiness questionnaire (PARQ), adverse reaction to BioFreeze, and body composition (hydrostatic weigh, bioelectrical impedance). Visits 2 and 3 will be separated by 7-14 days, randomized, and counterbalanced for experimental (BioFreeze) and control (hypoallergenic cream) trials. Both the experimental and control visits will follow the same protocol.

Participants will arrive following an overnight fast state while also refraining from strenuous activity, alcohol consumption, tobacco use, and recreational drugs for the previous 24 hour period. During these visit researchers will apply BioFreeze using a gloved hand from shoulder to wrist and mid thigh to ankle (areas outside of the clothing). A hypoallergenic cream will be applied during the control visit.

Exercise will consist of 30 min of moderate intensity treadmill walking (3.5 mph at 5% grade) within a heated temperature/humidity controlled chamber (38°C, 60% relative humidity). Participants will be weighed before, and after completion of the exercise calculate sweat rate. Prior to the exercise session, participants will sit for 5 min in an ambient room temperature environment as a baseline. During baseline and during the exercise core temperature, skin temperature, laser doppler blood flow, galvanic skin response, and heart rate will be collected continuously. Sweat patches will be adhered to the forehead during exercise at minute 10 for collection of sweat composition over the next 10-20 minutes. Thermal perception using the ASHRAE scale (cold to hot) will be assessed pre and during exercise.

VISIT 1 Visit 1 will take approximately 1 hour. Informed consent will be given. Participants will then complete the physical activity readiness questionnaire (PARQ) to be cleared for physical activity. Participants will have a small amount of the BioFreeze cream applied to a small area of the forearm (~2 x 2 in) to test for any adverse reaction over a period of 15 minutes. This initial skin reaction test is not a part of the research protocol. Those without a reaction will have height, weight, and body fat composition measured. Height and weight will be measured using a medical scale and stadiometer, respectively. Body fat will be assessed with hydrostatic weighing using an electronic load cell based system (Exertech, Dresbach, MN) correcting for residual lung volume or via a bio-electrical impedance analyzer (InBodyUSA, Cerritos, CA).

VISITS 2 AND 3 Visits 2 and 3 will take approximately 2 hours each. Upon arrival at the lab, a nude body weight will be collected with the subject in a private room. While still in the room, subjects will self-insert a rectal thermistor 12-15 cm beyond the anal sphincter and don a chest strap heart rate monitor. After dressing in their exercise clothing, subjects will exit the private room so that chest, forearm, and calf thermistors can be adhered to the skin with tape. Laser doppler flow (forearm and or/finger) will be adhered with tape and galvanic skin response (fingers) will be adhered using Velcro straps to the skin. Measuring instruments will be recorded using an integrated digital to analog converter (ADInstruments, Colorado Springs, CO).

Following instrumentation, subjects will sit for 5 minutes as a baseline in a temperate environment. Immediately after, a researcher with gloved hands will topically apply BioFreeze or the control hypoallergenic cream from the shoulder to wrist and mid-thigh to ankle. Subjects will then enter the heat chamber (38°C, 60% relative humidity) and immediately begin a 30-minute walk on a treadmill (3.5 mph, 5% grade). Subjects will be intermittently asked to hold their arm steady for laser doppler flow collection (10, 20, 30 minutes). Subjects will also briefly pause at minute 10 in order to adhere an absorbent patch to their forehead for sweat collection over the following 10-20 minutes. Thermal perception using the ASHRAE scale (cold to hot) will be assessed pre and during exercise. After 30 minutes of walking, subjects will exit the chamber for removal of all skin and finger sensors. Subjects will then re-enter the private room, remove their own rectal thermistor with gloved hands, and then a final nude body weight will be recorded after toweling off.

The rectal thermistor will measure core temperature. The heart rate monitor will measure the beats of the heart. Skin thermistors will measure the temperature of the skin surfaces. Laser doppler flow measure the relative units of blood flow velocity. Galvanic skin response measures skin conductivity changes as individuals begin to sweat. Sweat is collected for assessment of sweat composition. Thermal perception is assessed for individual perception surrounding the temperature of the ambient environment. Nude body weight is measured to calculate sweat rate.

ELIGIBILITY:
Inclusion Criteria:

* 19-45 years of age
* cleared for physical activity via the 2022 physical activity readiness questionnaire (PARQ)
* no self-reported adverse reactions to menthol based gels

Exclusion Criteria:

* outside 19-45 years of age
* not cleared for physical activity via the 2022 physical activity readiness questionnaire (PARQ)
* self-report or signs of sensitivity to menthol gels
* pregnant
* breast feeding

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin R Slivka, PhD, Principal Investigator — University of Montana
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Menthol Gel First, Then Hypoallergenic Gel: Participants randomized to receive menthol gel first then hypoallergenic gel after 7 day washout.
  All subjects complete both menthol gel and hypoallergenic gel conditions in a randomized cross-over study design. At least 7 days were allowed between conditions (washout).
  Menthol Gel: application of 5% menthol gel from shoulder to wrist and mid thigh to ankle
  Control Gel: application of hypoallergenic gel from shoulder to wrist and mid thigh to ankle
  Exercise: treadmill walking 3.5 mph at 5% grade
- Hypoallergenic Gel First, Then Menthol: Participants randomized to receive hypoallergenic gel first then menthol gel after 7 day washout.
  All subjects complete both menthol gel and hypoallergenic gel conditions in a randomized cross-over study design. At least 7 days were allowed between conditions (washout).
  Menthol Gel: application of 5% menthol gel from shoulder to wrist and mid thigh to ankle
  Control Gel: application of hypoallergenic gel from shoulder to wrist and mid thigh to ankle
  Exercise: treadmill walking 3.5 mph at 5% grade
Period: Overall Study
Arm/Group | Menthol Gel First, Then Hypoallergenic Gel | Hypoallergenic Gel First, Then Menthol
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Menthol gel will be applied to the skin or a A hypoallergenic gel will be applied to the skin prior to exercise in the heat.
  All subjects complete both menthol gel and hypoallergenic gel conditions in a randomized cross-over study design. At least 7 days were allowed between conditions (washout).
  Menthol Gel: application of 5% menthol gel from shoulder to wrist and mid thigh to ankle
  Control Gel: application of hypoallergenic gel from shoulder to wrist and mid thigh to ankle
  Exercise: treadmill walking 3.5 mph at 5% grade
  A hypoallergenic gel will be applied to the skin prior to exercise in the heat
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12
Body Composition [Mean (Standard Deviation); unit: percent body fat] | 20.1 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Skin Blood Flow
Description: Laser Doppler measurement of skin blood flow
Time Frame: 10 minutes into exercise bout
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Menthol Gel: Menthol Gel: application of 5% menthol gel from shoulder to wrist and mid thigh to ankle
  Menthol gel will be applied to the skin or a A hypoallergenic gel will be applied to the skin prior to exercise in the heat.
  All subjects complete both menthol gel and hypoallergenic gel conditions in a randomized cross-over study design. At least 7 days were allowed between conditions (washout).
  Exercise: treadmill walking 3.5 mph at 5% grade
- Control Gel: Control Gel: application of hypoallergenic gel from shoulder to wrist and mid thigh to ankle
  Menthol gel will be applied to the skin or a A hypoallergenic control gel will be applied to the skin prior to exercise in the heat.
  All subjects complete both menthol gel and hypoallergenic control gel conditions in a randomized cross-over study design. At least 7 days were allowed between conditions (washout).
  Exercise: treadmill walking 3.5 mph at 5% grade
Arm/Group | Menthol Gel | Control Gel
Number analyzed (Participants) | 12 | 12
arbitrary units | 131.6 (71.6) | 119.2 (43.2)
Statistical Analysis 1: Comparison: Menthol Gel vs Control Gel; Null hypothesis was there was no difference between menthol gel and control gel time x trial ANOVA statistical analysis; Test type: Superiority; p = 0.742, ANOVA — p-value reflects main effect of treatment

2. Primary Outcome: Skin Blood Flow
Description: Laser Doppler measurement of skin blood flow
Time Frame: 30 minutes into exercise bout
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Menthol: Menthol Gel: application of 5% menthol gel from shoulder to wrist and mid thigh to ankle
  Menthol gel will be applied to the skin or a A hypoallergenic gel will be applied to the skin prior to exercise in the heat. All subjects complete both menthol gel and hypoallergenic gel conditions in a randomized cross-over study design. At least 7 days were allowed between conditions (washout).
  Exercise: treadmill walking 3.5 mph at 5% grade
- Control: Control Gel: application of hypoallergenic gel from shoulder to wrist and mid thigh to ankle
  Menthol gel will be applied to the skin or a A hypoallergenic control gel will be applied to the skin prior to exercise in the heat. All subjects complete both menthol gel and hypoallergenic control gel conditions in a randomized cross-over study design. At least 7 days were allowed between conditions (washout).
  Exercise: treadmill walking 3.5 mph at 5% grade
Arm/Group | Menthol | Control
Number analyzed (Participants) | 12 | 12
arbitrary units | 196.1 (69.4) | 194.8 (73.3)
Statistical Analysis 1: Comparison: Menthol vs Control; The null hypothesis is that there is no difference between menthol and control trials; Test type: Superiority; p = 0.742, ANOVA — p-value is main effect of menthol

3. Primary Outcome: Galvanic Skin Response
Description: measurement of skin conductance
Time Frame: Time to 40 micro-siemens
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Menthol | Control
Number analyzed (Participants) | 12 | 12
seconds | 1299 (335) | 1148 (298)
Statistical Analysis 1: Comparison: Menthol vs Control; The null hypothesis is that there is no difference between menthol and control trials; Test type: Superiority; p = 0.048, ANOVA — p-value reflects main effect of menthol

4. Primary Outcome: Sweat Composition
Description: Sodium concentrations in collected sweat
Time Frame: final 10 minutes of exercise bout
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Menthol | Control
Number analyzed (Participants) | 12 | 12
mmol/L | 38.9 (13.8) | 43.9 (6.9)
Statistical Analysis 1: Comparison: Menthol vs Control; The null hypothesis is that there is no difference between menthol and control trials; Test type: Superiority; p = .104, t-test, 2 sided

5. Primary Outcome: Sweat Rate
Description: Difference in Nude body weight from pre to post exercise is assumed to be the amount of weight lost via sweat. This value is then expressed as liters of sweat lost per hour if the intervention was to last 1 hr.
Time Frame: pre to post exercise, approximately 30 minutes
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Menthol | Control
Number analyzed (Participants) | 12 | 12
Liters per hour | 1.1 (0.4) | 1.3 (.4)
Statistical Analysis 1: Comparison: Menthol vs Control; The null hypothesis is that there is no difference between menthol and control trials; Test type: Superiority; p = .051, t-test, 2 sided

6. Primary Outcome: Thermal Perception
Description: scale of thermal comfort developed by the American Society of Heating, Refrigerating and Air-Conditioning Engineers (ASHRAE). The ASHRAE is a 7-point scale to asses thermal sensation, which consists of seven verbal anchors: "cold (-3)", "cool (-2)", "slightly cool (-1)", "neutral (0)", "slightly warm (1)", "warm (2)", and "hot (3)". The score is reported as the value in "()"
Time Frame: throughout the 30 minute exercise bout
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Menthol | Control
Number analyzed (Participants) | 12 | 12
units on a scale | 0.7 (1.6) | 1.8 (1.3)
Statistical Analysis 1: Comparison: Menthol vs Control; The null hypothesis is that there is no difference between menthol and control trials; Test type: Superiority; p < 0.001, ANOVA — Main effect of treatment

7. Primary Outcome: Average Skin Temperature
Description: average measurements from chest, forearm, and calf thermistors
Time Frame: after 30 minutes of exercise
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Menthol | Control
Number analyzed (Participants) | 12 | 12
degrees C | 37.6 (.3) | 37.2 (.5)
Statistical Analysis 1: Comparison: Menthol vs Control; The null hypothesis is that there is no difference between menthol and control trials; Test type: Superiority; p = .026, ANOVA

8. Primary Outcome: Core Temperature
Description: measured with rectal thermistor
Time Frame: after 30min exercise
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Menthol | Control
Number analyzed (Participants) | 12 | 12
degrees C | 38.1 (.3) | 37.7 (.3)
Statistical Analysis 1: Comparison: Menthol vs Control; The null hypothesis is that there is no difference between menthol and control trials; Test type: Superiority; p = .001, ANOVA — p-value at time 30 min of exercise

9. Primary Outcome: Sweat Potassium Concentration
Description: this is a measure of the amount of potassium in the sweat
Time Frame: final 10 minutes of the exercise bout
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Menthol Gel | Control Gel
Number analyzed (Participants) | 12 | 12
mmol/L | 7.1 (1.2) | 6.9 (1.7)
Statistical Analysis 1: Comparison: Menthol Gel vs Control Gel; Test type: Superiority; p > 0.05, t-test, 2 sided

10. Secondary Outcome: % Body Fat
Description: this is a descriptive measure of the amount of total body weight that is fat. expressed as a percentage. Since this is a repeated measures study (each subject completed all conditions) this test was only done once before the experimental trials.
Time Frame: preliminary testing before beginning the study
Population: There is only 1 arm for this variable since it is descriptive of the total subjects that subsequently participate in each condition (repeated-measures).
Measure: Mean (Standard Deviation); unit: percent body fat
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
percent body fat | 20.1 (6.3)

11. Secondary Outcome: Skin Surface Area
Description: as for outcome 10
Time Frame: preliminary testing completed prior to the study procedures
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: meters squared
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
meters squared | 1.98 (.31)

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 1 month
Description: There was not substantial risk for serious adverse events or all-cause mortality
Groups:
- Menthol Gel Application: Menthol gel will be applied to the skin prior to exercise in the heat
  Hot environment: 38°C, 60% relative humidity
  Menthol Gel: application of 5% menthol gel from shoulder to wrist and mid thigh to ankle
  Exercise: treadmill walking 3.5 mph at 5% grade
- Hypoallergenic Gel Application: A hypoallergenic gel will be applied to the skin prior to exercise in the heat
  Hot environment: 38°C, 60% relative humidity
  Control Gel: application of hypoallergenic gel from shoulder to wrist and mid thigh to ankle
  Exercise: treadmill walking 3.5 mph at 5% grade
Arm/Group | Menthol Gel Application | Hypoallergenic Gel Application
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT05302804/Prot_SAP_001.pdf